CLINICAL TRIAL: NCT00002038
Title: Non-Comparative Study of Fluconazole in Patients With Serious Mycoses and Who Cannot Be Treated With Conventional Antifungal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 012C; 056-152
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-06

CONDITIONS: Candidiasis; Mycoses; HIV Infections
Keywords: Mycoses; Drugs, Investigational; Fluconazole
MeSH Terms: conditions — Candidiasis; Mycoses; HIV Infections | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
The primary purpose of this protocol is to provide fluconazole for the treatment of individual patients who require therapy for serious or life-threatening systemic fungal infection, who have failed on conventional antifungal therapy or have had unacceptable reactions to conventional antifungal therapy, and who are ineligible for other established fluconazole clinical trial protocols.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

A patient will be excluded if he/she has previously had an unacceptable adverse effect due to fluconazole.

A patient will be excluded if he/she has previously had an unacceptable adverse effect due to fluconazole.

AMENDED:

* 900207 Open only to unapproved indications and/or age ranges.
* Original design:
* Patients with clinically established serious or life-threatening systemic fungal disease will be considered if conventional fungal therapy is not an acceptable alternative. Unacceptability of conventional therapy is defined as:
* Failure of conventional therapy to control or eradicate infection after appropriate trial(s) of generally accepted regimen(s).
* Serious and unacceptable untoward reaction(s) to conventional antifungal therapy.
* OR A major contraindication to the use of conventional antifungal therapy.
* The patient must be ineligible or have no access to other established fluconazole investigational protocols. The final judgment of patient acceptability for inclusion lies with the Pfizer Clinical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Pfizer Central Research, Groton, Connecticut, United States